CLINICAL TRIAL: NCT04257097
Title: Reinforced PTFE Meshes Versus Customized Titanium Meshes: Randomized Clinical Trial
Brief Title: Reinforced PTFE Meshes Versus Customized Titanium Meshes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GBR Academy (Network)
Responsible Party: Principal Investigator, Alessandro Cucchi, Principal Investigator, GBR Academy
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMF 01/2019
Record Dates: First submitted 2019-12-06; First posted 2020-02-05 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Surgical Procedure, Unspecified; Soft Tissue Infections; Surgical Wound Dehiscence; Bone Density; Bone Loss; Dental Implant Failed
MeSH Terms: conditions — Soft Tissue Infections; Surgical Wound Dehiscence; Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The surgeon is masked until the envelope is opened at the time of the surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A - control group (Active Comparator): 25 patients will undergo bone regeneration with a titanium reinforced PTFE Mesh (RPM - Osteogenics Lubbock Texas USA), manually shaped and modeled by the operator during surgery (traditional technique), covered with collagen membranes of medium-rapid resorption (Vitala - Osteogenics Lubbock Texas USA)
  Interventions: Device: RPM - Osteogenics Lubbock Texas USA
- Group B - Test group (Experimental): 25 patients undergo bone regeneration with a custom-made titanium mesh (Yxoss CBR - Reoss Filderstadt Germany), digitally designed by an operator before the surgery (digital technique), covered by collagen membranes with medium-rapid resorption (Bio-Gide - Geistlich Baden Baden Germany)
  Interventions: Device: Yxoss CBR - Reoss Filderstadt Germany

INTERVENTIONS:
Device: RPM - Osteogenics Lubbock Texas USA — 25 patients will undergo bone regeneration with a reinforced PTFE mesh, manually shaped and modelled by the operator during surgery (traditional technique), covered with collagen membranes of medium-rapid resorption
  Other Names: Vitala - Osteogenics Lubbock Texas USA
  Arms: Group A - control group
Device: Yxoss CBR - Reoss Filderstadt Germany — 25 patients undergo bone regeneration with a custom-made titanium mesh, digitally designed by an operator before the surgery (digital technique), covered by collagen membranes with medium-rapid resorption
  Other Names: Bio-Gide - Geistlich Baden Baden Germany
  Arms: Group B - Test group

SUMMARY:
The objective of this study is to compare two surgical techniques for the treatment of the maxillary and mandibular bone atrophies.. Therefore, the main purpose is to compare the (i) the percentage of post-operative complications (ii) the three-dimensional bone gain with customized titanium meshes (test group - the medical device is digitally designed and made with customized laser sintering modality, customized to the defect of each patient) and with titanium-reinforced PTFE mesh (control group - the medical device is cut, shaped, and manually modelled to the patient's defect by the operator himself.

DETAILED DESCRIPTION:
The rationale of the study is based on the fact that manual intra-operative modelling of a titanium-reinforced PTFE mesh is operator-dependent, and even in the case of very experienced operators it is always difficult, inaccurate and slow. The use of pre-modelled and pre-fabricated custom-made meshes with bevel margins and three-dimensional morphology adapted to the bone defect, would make it possible to carry out an important bone regeneration as it reduces the operating times, the risks linked to mesh borders, trauma to the soft tissues and the discomfort for the patient.

This study aims to evaluate, in cases of maxillary and mandibular atrophies characterized by a vertical and / or combined resorption of the alveolar bone, the complication rate (intra- and post-operative) and the three-dimensional bone gain after traditional bone regeneration, where the medical device necessary for bone regeneration is cut out, shaped, and manually modelled by the operator, compared to digital bone regeneration. Subsequently, the medical device is digitally designed and made with a computerized method.

The primary objective of the study is, therefore, the evaluation of the healing complications; in particular, the early or delayed exposure of medical devices used for bone regeneration, during the healing period. This exposure is, as reported in all clinical studies, the main cause of the failure of the surgery.

A secondary objective, is the quantitative assessment of bone regeneration obtained by the 2 techniques. In particular, the evaluation of the reconstructed bone volume (RBV) with respect to the planned bone volume (PBV).

Other targets include the qualitative evaluation of bone regeneration through histological and histomorphometric analysis of the bone biopsies obtained at the moment that the medical device is removed and finally the evaluation of the peri-implant bone resorption will be conducted over time.

This clinical trial, which is promoted by Prof. Giuseppe Corinaldesi and the Department of Biomedical and Neuromotor Sciences (DIBINEM), University of Bologna, is designed as a pilot, randomized, multicentric, independent, parallel-group clinical trial, in which the all variables will be analysed prospectively.

The study will have a selection and enrolment period of approximately 12 months and a treatment period of approximately 24 months. As a result, the overall duration of the study will be approximately 36 months.

Over the three-year period 2019/2021, it will include the treatment of 50 patients in good general health conditions who are affected by partial edentulism of the maxilla or mandible with vertical and horizontal resorption of the alveolar bone, which requires a prosthetic rehabilitation supported by implants to improve function and aesthetics of edentulous areas.

Patients will be divided into 2 study groups, according to the previously computer-generated randomization sequence the following will be assigned to each group: group A (control), 25 patients who will be treated with bone regeneration with titanium-reinforced PTFE mesh, shaped and manually modelled by the operator during surgery; group B (test), 25 patients will be treated with bone regeneration with titanium mesh, designed and produced before surgery.

The study will include 3 different treatment phases: the first phase (T0) involves bone regeneration using a standard technique (group A) or digital technique (group B); the second one (T1), subsequently, after 6 months, this will forsee the removal of the regeneration devices and the insertion of the implants; the third (T2), 3 months after the aforementioned, will forsee the final functional loading of the implants, with a consequent follow-up of the regenerated bone.

All the materials and tools that will be used in the study are CE certified (with the exception of the custom-made mesh which, as a custom-made device, does not require CE certification) and have already been used in the normal care path for patients who have undergone bone regeneration. Moreover, the control visits and the radiological investigations of the data foreseen by the aforementioned protocol will be collected; They will be summarized in the case report form (CRF), and are those that characterize the normal care path of patients undergoing necessary bone regeneration for prosthetic implant rehabilitation when the bone quantity is insufficient.

The primary objective of this study is to evaluate the non-inferiority of technique B (digital technique) compared to technique A (traditional technique) in the incidence of complications.

The Secondary objectives include: assessment of patient and operator benefits, reconstructed bone volume (RBV) compared to planned bone volume (PBV), histological and histomorphometric analysis of bone quality obtained and peri-implant bone resorption after 12 months of follow-up.

The sample size necessary to support the null hypothesis is 17 subjects for each group. In order to compensate for any protocol deviations or possible drop-outs, the number of patients was increased to 25 per group.

The results obtained in the two study groups will be subjected to descriptive statistical analysis and the differences between groups will be tested by means of appropriate statistical tests for purely exploratory and non-demonstrative purposes.

The patient will be considered as the statistical unit of the analysis, and the statistical significance will be set at α = 0.05.

The collected data will be grouped and summarized with respect to the demographic, anamnestic, and clinical variables of each patient.

Exploratory analyses will be performed using descriptive statistics. The data will be presented both for the intent-to-treat population and for the per-protocol population.

The sample size necessary to support the null hypothesis is 17 subjects for each group. In order to compensate for any protocol deviations or possible drop-outs, the number of patients was increased to 25 per group. The sample size was calculated using dedicated statistical software (STATA, StataCorp LLC) through Pearson's chi-squared test, guaranteeing a level of significance of 95% and a power of 80%.

ELIGIBILITY:
Inclusion Criteria:

Adult patients, over the age of 18, in good general health.

* Patients with partial edentulism of the maxilla or mandible, with a 2mm minimum to a 12mm maximum vertical bone defect, which requires a three-dimensional bone regeneration intervention in order to have a fixed implant supported rehabilitation.
* Obtaining informed consent for experimental treatment and processing the personal data.

Exclusion Criteria:

* Poor oral hygiene,

  * Untreated periodontal disease
  * Smoking habit> 10 cigarettes / day;
  * Abuse of alcohol or drugs
  * Pregnancy
  * Patients with odontostomatological infections and / or systemic infections in progress;
  * Patient with uncontrolled diabetes mellitus or other metabolic diseases;
  * Patients with severe changes in liver and kidney function.
  * Patients with confirmed uncontrolled autoimmune disorders.
  * Patients subjected radiation therapy in the head or neck region in the last 5 years.
  * Patients undergoing immunosuppressive and / or immunocompromised therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
The rate of healing complications after reconstructive surgery | 6 months
  Healing complications are evaluated based on the chronological order in which they occur:
  * immediate exposure occurs within the 1st month
  * early exposure occurs between the 1st and the 3rd month
  * late exposure occurs between after the 3rd month
  Evaluation of low-grade and high-grade infection of medical devices used for bone regeneration.
  The former complications are classified as:
  * Class A, including flap damage (soft tissue perforation or laceration)
  * Class B, including neurological damage (paresthesia or disesthesia)
  * Class C,including vascular damage (hemorrhage).
  The latter complications are divided into four classes, according to the presence and extent of exposure, as well as the presence of a purulent exudate:
  * Class I, membrane exposure <3 mm, no purulent exudate
  * Class II membrane exposure >=3mm, no purulent exudate
  * Class III: membrane exposure, with purulent exudate

SECONDARY OUTCOMES:
Level of anxiety of the patient measured with a Visual Analogue Scale (VAS) | Immediately before/after the surgery
  Level of anxiety measured with a Visual Analogue Scale (VAS), where 0 represents the absence of anxiety and 10 represents the maximum level of anxiety.
Pain level of the patient measured on a Visual Analogue Scale (VAS) | Post operative from immediately after surgery to the 14th day after the surgery.
  Pain level measured on a Visual Analogue Scale (VAS), where 0 represents the absence of pain and 10 represents the maximum level of pain.
Total Number of painkillers taken post-operative | Post operative from immediately after surgery to the 14th day after the surgery.
  Total amount of pain killers taken from post operative to the 14th day (a two week period) which will be recorded in the patient's diary.
Dosage of painkillers | Post operative from immediately after surgery to the 14th day after the surgery.
  Dosage of painkillers measured as the number of painkillers per day, which will be reported in a diary by the patients.
Limitation in daily functions measured on a Visual Analogue Scale (VAS) | Post operative from immediately after surgery to the 14th day after the surgery.
  Limitation in daily functions measured on a Visual Analogue Scale (VAS), where 0 represents the absence of limitations and 10 represents the total limitation
Number of patients' post-operative signs and symptoms | Post operative from immediately after surgery to the 14th day after the surgery.
  Self-assessment of patient's post-operative signs and symptoms (absence or presence swelling, nausea, hematoma, bruising, bleeding), which will be reported
Discomfort level of the patient using a Post-operative Symptom Severity (PoSSe) | Post operative, measured on 14th day after the surgery
  Discomfort level measured using a Post-operative Symptom Severity (PoSSe) questionnaire.
  Questions are a forced choice, requiring the respondent to tick one box.
  The questions evaluate the discomfort level in different areas:
  * eating: ability to eat, ability to swallow, enjoyment of food, altered taste sensation
  * speech: voice affected, inability to open mouth, speech affected
  * sensation: tingling of lips or tongue, numbness of lips or tongue
  * appearance: bruising of face and/or neck, swelling of face and/or neck, life affected by appearance
  * pain: days of pain, pain controlled by painkillers, life affected by pain
  * sickness: days of nausea and vomiting, number of attacks of nausea and vomiting on worst day
  * interference with daily activities: interference with work/housework/daily activities, interference with leisure activities
Level of satisfaction of the patient using a Health-Related Quality of Life (HrQoL) | Post operative, 6 months and 12 months after the dental prosthesis dental prosthesis has been placed.
  Level of satisfaction measured using a Health-Related Quality of Life (HrQoL) questionnaire. Each of the questions are answered with the options of "I am quite satisfied, I'm satisfied, I have no idea, I am dissatisfied, and I am quite dissatisfied".
  The questions evaluate:
  * satisfaction with the overall treatment
  * chewing ability
  * cleaning of the prothesis
  * esthetics of the prothesis
  * speaking ability
Willingness of the patient to undergo the intervention recorded on a Visual Analogue Scale (VAS) | Post operative measured on the 7th day and on the 14th day.
  Willingness to undergo the intervention recorded on a Visual Analogue Scale (VAS), where 0 corresponds to "I will never undergo this type of surgery again" and 10 corresponds to "no problem repeating surgery if necessary".
Time required for the CBCT analysis and design of the medical device | Pre-operative, 2 weeks before the day of the surgery
  Time required for the CBCT analysis and design of the medical device measured in a total number of minutes.
Total operative time required for the surgery measured from immediately before to immediately after the surgery. | During procedure
  Total operative time measured from the time of incision to the end of the suture.
Total chair time measured from immediately before the surgery to immediately after the surgery. | During procedure
  Total chair time measured from the time the patient enters the surgery to the time the patient leaves the room
Level of operator satisfaction Measured on a 5 point scale | Immediately after the surgery
  Level of operator satisfaction rated on a 5-point scale, ranging from ''0=absolutely not satisfied'' to ''5 = absolutely satisfied''
Level of operator confidence with the technique | During procedure
  Confidence level with the technique used on a 5-point rating scale, ranging from "0=absolutely not confident" to " 5 = absolutely confident"
Costs related to the technique | Immediately after surgery
  Costs related to the GBR technique measured as the total costs of the materials used: number of pins, number of screws, number of membranes, number of biomaterials, number of sutures
Operator anxiety level recorded on a Visual Analogue Scale (VAS) | From 3 days before the surgery to immediately before the surgery, during the intervention and at the 14th day after the surgery
  Operator anxiety level recorded on a Visual Analogue Scale (VAS), where 0 represents the absence of anxiety and 10 represents the maximum level of anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Corinaldesi, MD,DDS,MS, Study Director — School of dentistry - University of Bologna
Locations (1):
- School of Dentistry - University of Bologna, Bologna, Italy, Italy

IPD SHARING:
Plan to Share IPD: Yes
Original articles in international journals
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From January 2021
Access Criteria: Access credentials to journal resources